CLINICAL TRIAL: NCT06512610
Title: Validation of the Use of the "ELN 2022" Risk Stratification System in HLA MENAFC Patients Newly Diagnosed With Acute Myeloid Leukemia
Brief Title: ELN 2022 in MENAFC ( Middle Eastern or North Coast of Africa ) Patients With Newly AML
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Hemato02
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Leukemia, Myeloid
MeSH Terms: conditions — Leukemia, Myeloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Middle Eastern or North Coast of Africa patients with newly AML: Validation and refinement of the 2022 European LeukemiaNet genetic risk stratification of acute myeloid leukemia in MENAFC patients
  Interventions: Other: Middle Eastern or North Coast of Africa patients with newly AML

INTERVENTIONS:
Other: Middle Eastern or North Coast of Africa patients with newly AML — Validation and refinement of the 2022 European LeukemiaNet genetic risk stratification of acute myeloid leukemia in MENAFC patients
  Other Names: No treatment intervention. Evaluation of the European leukemia net 2022 classification.

SUMMARY:
"In daily clinical practice, 2022 ELN guidelines were used to predict response to conventional treatment and to guide the need for allogenic stem cell transplantation. But, the team has to underline that ELN guidelines are mainly reflective of relatively young Caucasian patients. Few studies have compared 2017 and 2022 ELN in ethnicity cohorts to evaluate the potential prognostic value of this new criteria in these types of population. For example, with the 2022 ELN guidelines, the disease-free surviva) and the overall survival of African American < 60 y.o were not statistically different between intermediate and adverse groups (p=0.30, p=0,46). There were not a significant difference between favorable and intermediate groups in DFS (p=0.42, p=0.42) respectively in African American and Hispanic patients or in OS (p=0.67) in Hispanic patients. Is the 2022 ELN applicable to all ethnic subgroups? To date, no studies have examined and validated its applicability in Middle Eastern or North Coast of Africa (MENAFC) patients."

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML
* At least 18 yo
* MENAFC (Middle East ern of North Coast of Africa) patients with HLA HLA > 50%
* ECOG performance status of 0,1,2,3"

Exclusion Criteria:

* Acute promyelocytic leukemia
* Patients alive at the start of the study who did not receive study information or who objected to the collection of data"

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HLA, Middle Eastern or North Coast of Africa, acute myeloid leukemia patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival according to ELN 2022 genetic-risk group in comparison to ELN 2017 | Time from first administration of induction chemotherapy to death from any cause, assessed up to 01/01/2025
  Patient alive or not. Patient alive at last follow-up were censored.

SECONDARY OUTCOMES:
Relapse free survival before alloHSCT | Time from date of complete remission to date of relapse or death from any cause, assessed up to 01/01/2025
  Patient who relapsed (confirmation with bone marow sample or MRD + Minimum residual Disease) / who died from any cause during the follow-up or patient with complete remission.
Risk group according to 2017 and 2022 ELN | At the diagnosis
  Presence of genetic abnormalities resulting in 3 risks categories: favorable, Intermediate and Adverse
Complete remission rates | Time from first administration of induction chemotherapy to death from any cause, assessed up to 01/01/2025
  complete remission rates %
Safety and tolerance | Time from first administration of induction chemotherapy to death from any cause, assessed up to 01/01/2025
  "Number of chemotherapy-related adverse events. Adverse events (AEs) were evaluated according to Common Terminology Criteria for Adverse Events classification: CTCAE (Version 4.0). Grade 1 = Mild - transient or mild discomfort; no limitation in activity; no medical intervention/therapy required
  * Grade 2 = Moderate - mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention/therapy required
  * Grade 3 = Severe - marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalization is possible
  * Grade 4 = Life threatening - extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable
  * Grade 5 = Death "

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France